CLINICAL TRIAL: NCT00443300
Title: Effectiveness of HEPA-filtered Rooms ("Protected Environment") to Prevent Morbidity and Mortality in Patients Age >/ = 60 Receiving Lower Intensity ("Targeted") Therapy for Untreated AML and High-risk Myelodysplasia (MDS)
Brief Title: Effectiveness of Protected Environment Rooms for AML and MDS
Status: Terminated | Type: Observational
Why Stopped: Terminated due to low accrual.
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2006-0696
Record Dates: First submitted 2007-03-01; First posted 2007-03-05 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-08

CONDITIONS: Acute Myelogenous Leukemia; Myelodysplastic Syndrome
Keywords: AML; MDS; Protected Environment
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Protective environment: Participants in a Protective environment
- Not a protective environment: Participants not in a protective environment

SUMMARY:
The goal of this clinical research study is to learn if the "protected environment" (PE) can help to prevent infections in patients aged 60 and above who are receiving what is considered low-intensity treatment for newly-diagnosed AML or high-risk MDS.

DETAILED DESCRIPTION:
For AML or high-risk MDS, it has been common practice for patients aged 50 and older to receive initial treatment in the PE at M. D. Anderson. The PE is a series of rooms containing a special air-flow system that is designed to filter out germs that can cause serious infection. Patients stay in a PE room, without leaving, for up to 5 weeks. In an attempt to keep a PE room germ-free, only the medical staff is allowed in the room. Family and visitors can see the patient, but are separated from the patient by a glass wall. Each PE room has a laptop computer that can be connected to the internet. Books, newspapers, and various other materials are only allowed in the PE room after they have been sterilized for safety reasons.

Therapy given to patients with AML or MDS has recently changed from higher (which usually meant that there was more possibility for infections and a need for hospitalization) to lower intensity. Because the value of the PE was already established in patients receiving higher-intensity therapy, researchers want to learn about the value of the PE in patients receiving lower-intensity therapy.

If you agree to take part in this study, you will be randomly assigned (as in the flip of a coin) to 1 of 2 groups. You will have an equal chance of being in either one of the groups. Participants in one group will be placed in the PE. Participants in the other group will not be placed in the PE but will have outpatient care. After the first 30 participants have been assigned to one group or the other, the chances of future participants being assigned to the PE will depend on the results (rates of infection) seen in earlier participants.

If you are assigned to the PE, you will stay in the PE for 5 weeks after beginning your standard treatment. You will be removed from the PE if medical problems develop that require you to receive treatment somewhere else in the hospital or if staying in the PE is simply too difficult (such as because of claustrophobia [fear of being in a closed space] or because of a feeling of "home sickness" [a strong desire to have physical contact with family and friends]).

If you are not assigned to the PE, you will be asked to stay in Houston for 5 weeks and will receive treatment on an outpatient basis, unless you have problems that require hospitalization (not in the PE).

You may choose not to be assigned to either group. If this is the case, the study doctor or study staff will ask you to participate in this study through allowing your data (information) to be collected.

If you choose not to be assigned and you agree, study staff will collect data regarding your rates of infections and remission (inactive disease) and the status of your health over time so that this information can be compared with rates seen in patients who took part in 1 of the 2 groups. This comparison information will be used to learn the value of the PE in patients receiving lower-intensity therapy. Up to 125 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

* AML or high-risk MDS (> 10% blasts in the marrow or blood)
* Patient is to be given "targeted therapy". Examples of targeted therapies are tipifarnib + low-dose ara-C, decitabine, and 5 azacitidine + valproic acid.
* Age >/= 60 years and Zubrod performance status of 0,1, or 2
* Informed consent obtained

Exclusion Criteria:

* Cannot receive ara-C at a dose >/= 100 mg/m2 daily, anthracyclines, or cloretazine.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with AML or high-risk MDS Age >/= 60 years with a Zubrod performance status of 0,1, or 2
Sampling Method: Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2007-01; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Success Rate | Baseline to 6 weeks post randomization to PE or Non PE
  Success is defined as number of participants with no death, pneumonia, or sepsis within 6 weeks of randomization compared to total number of participants to evaluate effect of the protected environment (PE) by (adaptively) randomly assigning patients age >/= 60 given targeted therapies between treatment inside or outside the PE.

CONTACTS AND LOCATIONS:
Overall Officials: Gloria N. Mattiuzzi, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M.D. Anderson's website — http://mdanderson.org